CLINICAL TRIAL: NCT01682837
Title: Value of Liquid Potassium Magnesium Citrate in Controlling Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LiqKMgCit-1208-01
Record Dates: First submitted 2012-09-04; First posted 2012-09-11 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (24):
- KMgCit, KCit, KCl, Placebo (Experimental): Participants who received study drug in the order: Potassium Magnesium Citrate (KMgCit) powder, Potassium Citrate (KCit) powder, Potassium Chloride (KCl) powder, Placebo. Study medications were taken twice daily after dissolution in 250 ml water. Each phase was followed by at least 1 week of washout.
  Interventions: Drug: Potassium chloride powder; Drug: Potassium citrate powder; Drug: Potassium magnesium citrate powder; Drug: Placebo
- KMgCit, KCit, Placebo, KCl (Experimental): Participants who received study drug in the order: Potassium Magnesium Citrate powder, Potassium Citrate powder, Placebo, Potassium Chloride powder. Study medications were taken twice daily after dissolution in 250 ml water. Each phase was followed by at least 1 week of washout.
  Interventions: Drug: Potassium chloride powder; Drug: Potassium citrate powder; Drug: Potassium magnesium citrate powder; Drug: Placebo
- KMgCit, KCl, KCit, Placebo (Experimental): Participants who received study drug in the order: Potassium Magnesium Citrate powder, Potassium Chloride powder, Potassium Citrate powder, Placebo. Study medications were taken twice daily after dissolution in 250 ml water. Each phase was followed by at least 1 week of washout.
  Interventions: Drug: Potassium chloride powder; Drug: Potassium citrate powder; Drug: Potassium magnesium citrate powder; Drug: Placebo
- KMgCit, KCl, Placebo, KCit (Experimental): Participants who received study drug in the order: Potassium Magnesium Citrate powder, Potassium Chloride powder, Placebo, Potassium Citrate powder. Study medications were taken twice daily after dissolution in 250 ml water. Each phase was followed by at least 1 week of washout.
  Interventions: Drug: Potassium chloride powder; Drug: Potassium citrate powder; Drug: Potassium magnesium citrate powder; Drug: Placebo
- KMgCit, Placebo, KCit, KCl (Experimental): Participants who received study drug in the order: Potassium Magnesium Citrate powder, Placebo, Potassium Citrate powder, Potassium Chloride powder. Study medications were taken twice daily after dissolution in 250 ml water. Each phase was followed by at least 1 week of washout.
  Interventions: Drug: Potassium chloride powder; Drug: Potassium citrate powder; Drug: Potassium magnesium citrate powder; Drug: Placebo
- KMgCit, Placebo, KCl, KCit (Experimental): Participants who received study drug in the order: Potassium Magnesium Citrate powder, Placebo, Potassium Chloride powder, Potassium Citrate powder. Study medications were taken twice daily after dissolution in 250 ml water. Each phase was followed by at least 1 week of washout.
  Interventions: Drug: Potassium chloride powder; Drug: Potassium citrate powder; Drug: Potassium magnesium citrate powder; Drug: Placebo
- KCit, KMgCit, KCl, Placebo (Experimental): Participants who received study drug in the order: Potassium Citrate powder, Potassium Magnesium Citrate powder, Potassium Chloride powder, Placebo. Study medications were taken twice daily after dissolution in 250 ml water. Each phase was followed by at least 1 week of washout.
  Interventions: Drug: Potassium chloride powder; Drug: Potassium citrate powder; Drug: Potassium magnesium citrate powder; Drug: Placebo
- KCit, KMgCit, Placebo, KCl (Experimental): Participants who received study drug in the order: Potassium Citrate powder, Potassium Magnesium Citrate powder, Placebo, Potassium Chloride powder. Study medications were taken twice daily after dissolution in 250 ml water. Each phase was followed by at least 1 week of washout.
  Interventions: Drug: Potassium chloride powder; Drug: Potassium citrate powder; Drug: Potassium magnesium citrate powder; Drug: Placebo
- KCit, KCl, KMgCit, Placebo (Experimental): Participants who received study drug in the order: Potassium Citrate powder, Potassium Chloride powder, Potassium Magnesium Citrate powder, Placebo. Study medications were taken twice daily after dissolution in 250 ml water. Each phase was followed by at least 1 week of washout.
  Interventions: Drug: Potassium chloride powder; Drug: Potassium citrate powder; Drug: Potassium magnesium citrate powder; Drug: Placebo
- KCit, KCl, Placebo, KMgCit (Experimental): Participants who received study drug in the order: Potassium Citrate powder, Potassium Chloride powder, Placebo, Potassium Magnesium Citrate powder. Study medications were taken twice daily after dissolution in 250 ml water. Each phase was followed by at least 1 week of washout.
  Interventions: Drug: Potassium chloride powder; Drug: Potassium citrate powder; Drug: Potassium magnesium citrate powder; Drug: Placebo
- KCit, Placebo, KMgCit, KCl (Experimental): Participants who received study drug in the order: Potassium Citrate powder, Placebo, Potassium Magnesium Citrate powder, Potassium Chloride powder. Study medications were taken twice daily after dissolution in 250 ml water. Each phase was followed by at least 1 week of washout.
  Interventions: Drug: Potassium chloride powder; Drug: Potassium citrate powder; Drug: Potassium magnesium citrate powder; Drug: Placebo
- KCit, Placebo, KCl, KMgCit (Experimental): Participants who received study drug in the order: Potassium Citrate powder, Placebo, Potassium Chloride powder, Potassium Magnesium Citrate powder. Study medications were taken twice daily after dissolution in 250 ml water. Each phase was followed by at least 1 week of washout.
  Interventions: Drug: Potassium chloride powder; Drug: Potassium citrate powder; Drug: Potassium magnesium citrate powder; Drug: Placebo
- KCl, KMgCit, KCit, Placebo (Experimental): Participants who received study drug in the order: Potassium Chloride powder, Potassium Magnesium Citrate powder, Potassium Citrate powder, Placebo. Study medications were taken twice daily after dissolution in 250 ml water. Each phase was followed by at least 1 week of washout.
  Interventions: Drug: Potassium chloride powder; Drug: Potassium citrate powder; Drug: Potassium magnesium citrate powder; Drug: Placebo
- KCl, KMgCit, Placebo, KCit (Experimental): Participants who received study drug in the order: Potassium Chloride powder, Potassium Magnesium Citrate powder, Placebo, Potassium Citrate powder. Study medications were taken twice daily after dissolution in 250 ml water. Each phase was followed by at least 1 week of washout.
  Interventions: Drug: Potassium chloride powder; Drug: Potassium citrate powder; Drug: Potassium magnesium citrate powder; Drug: Placebo
- KCl, KCit, KMgCit, Placebo (Experimental): Participants who received study drug in the order: Potassium Chloride powder, Potassium Citrate powder, Potassium Magnesium Citrate powder, Placebo. Study medications were taken twice daily after dissolution in 250 ml water. Each phase was followed by at least 1 week of washout.
  Interventions: Drug: Potassium chloride powder; Drug: Potassium citrate powder; Drug: Potassium magnesium citrate powder; Drug: Placebo
- KCl, KCit, Placebo, KMgCit (Experimental): Participants who received study drug in the order: Potassium Chloride powder, Potassium Citrate powder, Placebo, Potassium Magnesium Citrate powder. Study medications were taken twice daily after dissolution in 250 ml water. Each phase was followed by at least 1 week of washout.
  Interventions: Drug: Potassium chloride powder; Drug: Potassium citrate powder; Drug: Potassium magnesium citrate powder; Drug: Placebo
- KCl, Placebo, KMgCit, KCit (Experimental): Participants who received study drug in the order: Potassium Chloride powder, Placebo, Potassium Magnesium Citrate powder, Potassium Citrate powder. Study medications were taken twice daily after dissolution in 250 ml water. Each phase was followed by at least 1 week of washout.
  Interventions: Drug: Potassium chloride powder; Drug: Potassium citrate powder; Drug: Potassium magnesium citrate powder; Drug: Placebo
- KCl, Placebo, KCit, KMgCit (Experimental): Participants who received study drug in the order: Potassium Chloride powder, Placebo, Potassium Citrate powder, Potassium Magnesium Citrate powder. Study medications were taken twice daily after dissolution in 250 ml water. Each phase was followed by at least 1 week of washout.
  Interventions: Drug: Potassium chloride powder; Drug: Potassium citrate powder; Drug: Potassium magnesium citrate powder; Drug: Placebo
- Placebo, KMgCit, KCit, KCl (Experimental): Participants who received study drug in the order: Placebo, Potassium Magnesium Citrate powder, Potassium Citrate powder, Potassium Chloride powder. Study medications were taken twice daily after dissolution in 250 ml water. Each phase was followed by at least 1 week of washout.
  Interventions: Drug: Potassium chloride powder; Drug: Potassium citrate powder; Drug: Potassium magnesium citrate powder; Drug: Placebo
- Placebo, KMgCit, KCl, KCit (Experimental): Participants who received study drug in the order: Placebo, Potassium Magnesium Citrate powder, Potassium Chloride powder, Potassium Citrate powder. Study medications were taken twice daily after dissolution in 250 ml water. Each phase was followed by at least 1 week of washout.
  Interventions: Drug: Potassium chloride powder; Drug: Potassium citrate powder; Drug: Potassium magnesium citrate powder; Drug: Placebo
- Placebo, KCit, KMgCit, KCl (Experimental): Participants who received study drug in the order: Placebo, Potassium Citrate powder, Potassium Magnesium Citrate powder, Potassium Chloride powder. Study medications were taken twice daily after dissolution in 250 ml water. Each phase was followed by at least 1 week of washout.
  Interventions: Drug: Potassium chloride powder; Drug: Potassium citrate powder; Drug: Potassium magnesium citrate powder; Drug: Placebo
- Placebo, KCit, KCl, KMgCit (Experimental): Participants who received study drug in the order: Placebo, Potassium Citrate powder, Potassium Chloride powder, Potassium Magnesium Citrate powder. Study medications were taken twice daily after dissolution in 250 ml water. Each phase was followed by at least 1 week of washout.
  Interventions: Drug: Potassium chloride powder; Drug: Potassium citrate powder; Drug: Potassium magnesium citrate powder; Drug: Placebo
- Placebo, KCl, KMgCit, KCit (Experimental): Participants who received study drug in the order: Placebo, Potassium Chloride powder, Potassium Magnesium Citrate powder, Potassium Citrate powder. Study medications were taken twice daily after dissolution in 250 ml water. Each phase was followed by at least 1 week of washout.
  Interventions: Drug: Potassium chloride powder; Drug: Potassium citrate powder; Drug: Potassium magnesium citrate powder; Drug: Placebo
- Placebo, KCl, KCit, KMgCit (Experimental): Participants who received study drug in the order: Placebo, Potassium Chloride powder, Potassium Citrate powder, Potassium Magnesium Citrate powder. Study medications were taken twice daily after dissolution in 250 ml water. Each phase was followed by at least 1 week of washout.
  Interventions: Drug: Potassium chloride powder; Drug: Potassium citrate powder; Drug: Potassium magnesium citrate powder; Drug: Placebo

INTERVENTIONS:
Drug: Potassium chloride powder — 1 sachet mixed with 250 ml water (providing 20 meq K) given at breakfast and again dinner, for a total of 40 meq K/day, for 4 weeks
  Other Names: KCl
Drug: Potassium citrate powder — 1 sachet mixed with 250 ml water (providing 20 meq K) given at breakfast and dinner, for a total of 40 meq K/day, for 4 weeks
  Other Names: KCit
Drug: Potassium magnesium citrate powder — 1 sachet mixed with 250 ml water (providing 20 meq K) given at breakfast and dinner, for a total of 40 meq K/day, for 4 weeks
  Other Names: KMgCit
Drug: Placebo — 1 sachet mixed with 250 ml water given at breakfast and dinner, for a total of 2 sachets/day, for 4 weeks
  Other Names: Microcystalline cellulose

SUMMARY:
Liquid potassium-magnesium citrate (KMgCit) as a pharmaceutical formulation will lower blood pressure among patients with pre- or Stage I hypertension on their customary diet.

DETAILED DESCRIPTION:
In this protocol, the investigators want to explore whether KMgCit taken during a customary dietary setting, might serve as a "surrogate" for the Dietary Approaches to Stop Hypertension (DASH) diet to lower blood pressure. This study has obvious biomedical importance. Lifestyle modifications are often recommended for pre- or Stage I hypertension. The DASH diet is such a modification that has been shown to be effective. However, this diet is costly and difficult to adhere to long-term. If KMgCit were shown to be effective in lowering blood pressure, it would provide a safe and convenient alternative to the DASH diet.

ELIGIBILITY:
Inclusion Criteria:

* Men or women > 21 years of age
* Any Race/Ethnicity
* Pre- or Stage I hypertension (BP >= 120/80 and <= 159/99)

Exclusion Criteria:

* Diabetes mellitus
* Renal impairment (serum creatinine > 1.4 mg/dL)
* Any heart diseases such as congestive heart failure or sustained arrhythmia
* Chronic NSAID use
* Treatment with diuretics
* Gastroesophageal reflux disease (GERD) requiring treatment with acid reducing agents or antacid more than once a week
* Esophageal-gastric ulcer
* Chronic diarrhea
* Hyperkalemia (serum > 4.6 meq/L for patients on angiotension-converting-enzyme (ACE) inhibitors or angiotensin receptor blockers (ARBs), serum K > 5.0 meq/L for patient not on ACE inhibitors or ARBs)
* Abnormal liver function test (aspartate transaminase (AST) or alanine transaminase (ALT) above upper limit of normal range)
* Subjects who require any potassium supplement on a regular basis from any reasons
* Pregnancy
* History of major depression, bipolar disorder, or schizophrenia

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wanpen Vongpatanasin, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Hypertension Clinic - UT Southwestern Medical Center at Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vongpatanasin W, Peri-Okonny P, Velasco A, Arbique D, Wang Z, Ravikumar P, Adams-Huet B, Moe OW, Pak CYC. Effects of Potassium Magnesium Citrate Supplementation on 24-Hour Ambulatory Blood Pressure and Oxidative Stress Marker in Prehypertensive and Hypertensive Subjects. Am J Cardiol. 2016 Sep 15;118(6):849-853. doi: 10.1016/j.amjcard.2016.06.041. Epub 2016 Jun 28. PMID 27448942

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: Participants received the following study drug in random order: Potassium Magnesium Citrate (KMgCit) powder, Potassium Citrate (KCit) powder, Potassium Chloride (KCl) powder and Placebo. Study medications were taken twice daily after dissolution in 250 ml water. Each phase was followed by at least 1 week of washout. Individual study drug assignments per randomization is provided in the comments for each study period.
Period: Baseline
Arm/Group | All Study Participants
Started | 35
Completed | 30
Not Completed | 5
Not completed — Withdrawal by Subject | 5
Period: First Intervention (4 Weeks)
Arm/Group | All Study Participants
Started | 30
Received KMgCit | 8
Received KCit | 8
Received KCl | 7
Received Placebo | 7
Completed | 30
Not Completed | 0
Period: Second Intervention (4 Weeks)
Arm/Group | All Study Participants
Started | 30
Received KMgCit | 7
Received KCit | 6
Received KCl | 8
Received Placebo | 9
Completed | 30
Not Completed | 0
Period: Third Intervention (4 Weeks)
Arm/Group | All Study Participants
Started | 30
Received KMgCit | 9
Received KCit | 7
Received KCl | 7
Received Placebo | 7
Completed | 30
Not Completed | 0
Period: Fourth Intervention (4 Weeks)
Arm/Group | All Study Participants
Started | 30
Received KMgCit | 6
Received KCit | 9
Received KCl | 8
Received Placebo | 7
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Thirty (30) subjects participated in the trial. Each subject completed all four phases of the trial.
Groups:
- All Study Participants: Participants received the following study drug in random order: Potassium Magnesium Citrate powder, Potassium Citrate powder, Potassium Chloride powder, Placebo. Study medications were taken twice daily after dissolution in 250 ml water. Each phase was followed by at least 1 week of washout.
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31 (5)
Office Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 125 (11)
Office Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 81 (8)
Office Heart Rate [Mean (Standard Deviation); unit: beats per minute] | 72 (11)
24-hr Systolic Blood Pressure Average [Mean (Standard Deviation); unit: mmHg] | 126 (10)
24-hr Diastolic Blood Pressure Average [Mean (Standard Deviation); unit: mmHg] | 79 (10)
24-hr Heart Rate Average [Mean (Standard Deviation); unit: beats per minute] | 76 (11)
24-hr Daytime Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 129 (10)
24-hr Daytime Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 81 (11)
24-hr Daytime Heart Rate [Mean (Standard Deviation); unit: beats per minute] | 77 (11)
24-hr Nighttime Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 117 (12)
24-hr Nighttime Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 71 (10)
24-hr Nighttime Heart Rate [Mean (Standard Deviation); unit: beats per minute] | 70 (11)
Serum Calcium [Mean (Standard Deviation); unit: mg/dl] | 9.5 (0.5)
Serum Phosphorus [Mean (Standard Deviation); unit: mg/dl] | 3.6 (0.1)
Serum Magnesium [Mean (Standard Deviation); unit: mg/dl] | 2.2 (0.3)
Serum Sodium [Mean (Standard Deviation); unit: meq/L] | 139 (2)
Serum Potassium [Mean (Standard Deviation); unit: meq/L] | 4.2 (0.3)
Serum Chloride (meq/L) [Mean (Standard Deviation); unit: meq/L] | 105 (2)
Serum Bicarbonate [Mean (Standard Deviation); unit: meq/L] | 23 (2)
Serum Urea Nitrogen [Mean (Standard Deviation); unit: mg/dl] | 13.7 (3.5)
Serum Creatinine (mg/dl) [Mean (Standard Deviation); unit: mg/dl] | 0.9 (0.2)
Serum Albumin [Mean (Standard Deviation); unit: g/dl] | 4.2 (0.6)
Serum Parathyroid Hormone [Mean (Standard Deviation); unit: pg/ml] | 59 (31)
Serum 1,25-Dihydroxyvitamin D [Mean (Standard Deviation); unit: pg/ml] | 73 (34)

OUTCOME MEASURES:

1. Primary Outcome: 24-hour Average Systolic Blood Pressure
Description: This is the average systolic blood pressure over a 24 hour period.
Time Frame: 4 weeks
Population: All participants who completed the study completed all 4 phases.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Potassium Magnesium Citrate Powder Phase: Participants undergoing the Potassium Magnesium Citrate powder phase of the study.
- Potassium Citrate Powder Phase: Participants undergoing the Potassium Citrate powder phase of the study.
- Potassium Chloride Powder Phase: Participants undergoing the Potassium Chloride powder phase of the study.
- Placebo Phase: Participants undergoing the Placebo phase of the study.
Arm/Group | Potassium Magnesium Citrate Powder Phase | Potassium Citrate Powder Phase | Potassium Chloride Powder Phase | Placebo Phase
Number analyzed (Participants) | 30 | 30 | 30 | 30
mmHg | 127 (11) | 127 (10) | 126 (9) | 129 (13)
Statistical Analysis 1: Comparison: Potassium Magnesium Citrate Powder Phase vs Potassium Citrate Powder Phase vs Potassium Chloride Powder Phase vs Placebo Phase; Test type: Superiority or Other; p = 0.07, Mixed Models Analysis

2. Primary Outcome: 24-hour Average Diastolic Blood Pressure
Description: The average diastolic blood pressure over a 24 hour period.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Potassium Magnesium Citrate Powder Phase | Potassium Citrate Powder Phase | Potassium Chloride Powder Phase | Placebo Phase
Number analyzed (Participants) | 30 | 30 | 30 | 30
mmHg | 79 (10) | 78 (9) | 78 (9) | 80 (11)
Statistical Analysis 1: Comparison: Potassium Magnesium Citrate Powder Phase vs Potassium Citrate Powder Phase vs Potassium Chloride Powder Phase vs Placebo Phase; Test type: Superiority or Other; p = 0.20, Mixed Models Analysis

3. Secondary Outcome: Office Systolic Blood Pressure
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Potassium Magnesium Citrate Powder Phase | Potassium Citrate Powder Phase | Potassium Chloride Powder Phase | Placebo Phase
Number analyzed (Participants) | 30 | 30 | 30 | 30
mmHg | 124 (11) | 125 (13) | 127 (11) | 129 (12)
Statistical Analysis 1: Comparison: Potassium Magnesium Citrate Powder Phase vs Potassium Citrate Powder Phase vs Potassium Chloride Powder Phase vs Placebo Phase; Test type: Superiority or Other; p = 0.16, Mixed Models Analysis

4. Secondary Outcome: Office Diastolic Blood Pressure
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Potassium Magnesium Citrate Powder Phase | Potassium Citrate Powder Phase | Potassium Chloride Powder Phase | Placebo Phase
Number analyzed (Participants) | 30 | 30 | 30 | 30
mmHg | 81 (9) | 81 (8) | 80 (9) | 81 (9)
Statistical Analysis 1: Comparison: Potassium Magnesium Citrate Powder Phase vs Potassium Citrate Powder Phase vs Potassium Chloride Powder Phase vs Placebo Phase; Test type: Superiority or Other; p = 0.70, Mixed Models Analysis

5. Secondary Outcome: Serum C-terminal Telopeptide (CTX)
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Potassium Magnesium Citrate Powder Phase | Potassium Citrate Powder Phase | Potassium Chloride Powder Phase | Placebo Phase
Number analyzed (Participants) | 30 | 30 | 30 | 30
ng/ml | 0.46 (0.28) | 0.46 (0.28) | 0.45 (0.25) | 0.49 (0.33)
Statistical Analysis 1: Comparison: Potassium Magnesium Citrate Powder Phase vs Potassium Citrate Powder Phase vs Potassium Chloride Powder Phase vs Placebo Phase; Test type: Superiority or Other; p = 0.42, Mixed Models Analysis

6. Secondary Outcome: 24-hour Urinary Calcium
Time Frame: 4 weeks of treatment
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Potassium Magnesium Citrate Powder Phase | Potassium Citrate Powder Phase | Potassium Chloride Powder Phase | Placebo Phase
Number analyzed (Participants) | 30 | 30 | 30 | 30
mg/day | 158 (94) | 148 (78) | 160 (92) | 181 (101)
Statistical Analysis 1: Comparison: Potassium Magnesium Citrate Powder Phase vs Potassium Citrate Powder Phase vs Potassium Chloride Powder Phase vs Placebo Phase; Test type: Superiority or Other; p = 0.10, Mixed Models Analysis

7. Secondary Outcome: Carotid to Femoral Pulse Wave Velocity
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Potassium Magnesium Citrate Powder Phase | Potassium Citrate Powder Phase | Potassium Chloride Powder Phase | Placebo Phase
Number analyzed (Participants) | 30 | 30 | 30 | 30
m/s | 8.7 (1.7) | 8.8 (1.6) | 8.7 (1.5) | 8.9 (1.8)
Statistical Analysis 1: Comparison: Potassium Magnesium Citrate Powder Phase vs Potassium Citrate Powder Phase vs Potassium Chloride Powder Phase vs Placebo Phase; Test type: Superiority or Other; p = 0.64, Mixed Models Analysis

8. Secondary Outcome: Central Aortic Systolic Blood Pressure
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Potassium Magnesium Citrate Powder Phase | Potassium Citrate Powder Phase | Potassium Chloride Powder Phase | Placebo Phase
Number analyzed (Participants) | 30 | 30 | 30 | 30
mmHg | 121 (11) | 125 (16) | 123 (13) | 126 (14)
Statistical Analysis 1: Comparison: Potassium Magnesium Citrate Powder Phase vs Potassium Citrate Powder Phase vs Potassium Chloride Powder Phase vs Placebo Phase; Test type: Superiority or Other; p = 0.18, Mixed Models Analysis

9. Secondary Outcome: Central Aortic Diastolic Blood Pressure
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Potassium Magnesium Citrate Powder Phase | Potassium Citrate Powder Phase | Potassium Chloride Powder Phase | Placebo Phase
Number analyzed (Participants) | 30 | 30 | 30 | 30
mmHg | 77 (7) | 76 (7) | 77 (9) | 79 (8)
Statistical Analysis 1: Comparison: Potassium Magnesium Citrate Powder Phase vs Potassium Citrate Powder Phase vs Potassium Chloride Powder Phase vs Placebo Phase; Test type: Superiority or Other; p = 0.12, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during each subject's study period. Each study period was 4 weeks in duration.
Description: Systematic assessments were collected by a side effect questionaire which asked about Vomiting, Nausea, Belching, Diarrhea, Loose Bowel Movements, Pain/Cramp, Melena, Dyspepsia, Anorexia, Dysphagia, Dysgeusia and Other.
Arm/Group | Potassium Magnesium Citrate Powder Phase | Potassium Citrate Powder Phase | Potassium Chloride Powder Phase | Placebo Phase
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 5/30 | 5/30 | 16/30 | 4/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Potassium Magnesium Citrate Powder Phase (N=30) | Potassium Citrate Powder Phase (N=30) | Potassium Chloride Powder Phase (N=30) | Placebo Phase (N=30)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Belching (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Loose Bowel Movement (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (6) | 0 (0)
Pain and/or Cramps (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Gastrointestinal disorders) | 2 (3) | 2 (3) | 12 (18) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes